CLINICAL TRIAL: NCT05047978
Title: Growth and Tolerance of a Partially Hydrolyzed Cow's Milk Protein (PHP) Infant Formula
Brief Title: Growth and Tolerance of a Partially Hydrolyzed Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 3391-1
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Growth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A routine cow's milk-based infant formula (Active Comparator): A routine cow's milk-based infant formula
  Interventions: Other: Cow's milk protein infant formula
- A partially hydrolyzed cow's milk protein (PHP) infant formula (Experimental): A partially hydrolyzed cow's milk protein (PHP) infant formula
  Interventions: Other: Partially hydrolyzed protein infant formula

INTERVENTIONS:
Other: Cow's milk protein infant formula — A routine cow's milk-based infant formula
  Arms: A routine cow's milk-based infant formula
Other: Partially hydrolyzed protein infant formula — A partially hydrolyzed cow's milk protein (PHP) infant formula
  Arms: A partially hydrolyzed cow's milk protein (PHP) infant formula

SUMMARY:
The purpose of this research study is to compare the growth and tolerance of infants who consume either an infant formula with intact proteins or an infant formula with partially hydrolyzed proteins through approximately 12 months of age.

ELIGIBILITY:
Inclusion Criteria:

* 10 to 14 days of age at randomization
* singleton birth
* Gestational age of 37 to 42 weeks
* Birth weight of 2500 g (5lbs 8oz or more)
* Exclusively receiving infant formula for at least 24 hours prior to randomization
* Parent or legal guardian has full intention to exclusively feed study formula through 120 days of age
* Parent or legal guardian agrees not to enroll infant in another interventional clinical study while participating in this study
* Signed informed consent and authorization to use and disclose Protected Health information

Exclusion Criteria:

* History of underlying metabolic or chronic disease
* Evidence of feeding difficulties or history of formula intolerance
* Weight at Visit 1 is <98% of birth weight
* Infant was born large for gestational age from a mother who was diabetic at childbirth
* Infant is immunocompromised

Ages: 10 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 244 (Actual)
Dates: Start 2021-08-28 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Rate of body weight gain | up to 120 days

SECONDARY OUTCOMES:
Body length | up to 365 days of age
Head circumference | up to 365 days of age
Growth Z scores | up to 365 days of age
  weight-for-age
Growth Z scores | up to 365 days of age
  length-for-age
Growth Z scores | up to 365 days of age
  head circumference-for-age
Recall of study formula intake measured at each study visit | up to 365 days of age
  questionnaire
Recall of stool characteristics measured at each study visit | up to 365 days of age
  questionnaire
Pediatric Quality of Life Family Impact Module | up to 365 days of age
  questionnaire
Pediatric Quality of Life Inventory Infant Scales | 120, 180, 275, and 365 days of age
  Questionnaire. A 5-point response scale is utilized (0 = never a problem; 4 = always a problem). Items are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0), so that higher scores indicate better functioning (less negative impact).
Medically confirmed adverse events collected throughout the study period | up to 365 days of age
Specific medically confirmed adverse events related to gastrointestinal | up to 365 days of age
Specific medically confirmed adverse events related to allergy | up to 365 days of age
Body weight | up to 365 days of age

CONTACTS AND LOCATIONS:
Overall Officials: Steven Wu, Medical Director, Study Director — Mead Johnson Nutrition
Locations (13):
- United States (13):
  - Birmingham Pediatric Associates, Birmingham, Alabama
  - Southeastern Pediatric Associates, Dothan, Alabama
  - Visions Clinical Research-Tucson, Tucson, Arizona
  - Northwest Arkansas Pediatric Clinic, Fayetteville, Arkansas
  - The Children's Clinic of Jonesboro, Jonesboro, Arkansas
  - PAS Research, Tampa, Florida
  - Rophe Adult & Pediatric Medicine, Union City, Georgia
  - Saltzer Health, Nampa, Idaho
  - Springs Medical Research, Owensboro, Kentucky
  - Meridian Clinical Research, Grand Island, Nebraska
  - The Jackson Clinic, Jackson, Tennessee
  - DCOL Center for Clinical Research, Longview, Texas
  - PAS Research, McAllen, Texas

REFERENCES:
- [Derived] Fabrizio V, Abdelmagid SA, Bose A, Hale M, Hays EC, Hudson M, Hughes T, Leonard D, Rouse K, Sideri M, Walker J, Wampler JL, Yeiser M, Zhuang W, Wu SS. Partially hydrolyzed cow's milk protein formula with an added prebiotic is well-tolerated, safe, and supports age-appropriate growth in healthy term infants through one year of age: DBRCT. BMC Pediatr. 2026 Jan 13. doi: 10.1186/s12887-025-06454-2. Online ahead of print. PMID 41527066